CLINICAL TRIAL: NCT04745247
Title: Using a New Form of Cross-border Plasticity Within the Somatosensory Cortex: Stimulate the Face to Improve Tactile Acuity on the Hand
Brief Title: Stimulate the Face to Improve Tactile Acuity on the Hand
Acronym: FACEHAND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 69HCL20_0888; 2020-A03467-32 (Other: ID-RCB)
Record Dates: First submitted 2021-01-26; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Stroke; RSS; Face
MeSH Terms: conditions — Stroke; Facies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSS (Experimental): Repetitive somatosensory stimulation (RSS)
  Interventions: Procedure: RSS
- Sham RSS (Placebo Comparator): Sham Repetitive somatosensory stimulation (RSS)
  Interventions: Procedure: RSS

INTERVENTIONS:
Procedure: RSS — Repetitive somatosensory stimulation (RSS) applied on a small region of the face for 3 hours
  Sham Repetitive somatosensory stimulation (RSS) applied on a small region of the face for 3 hours : the number of stimuli is reduced compared to the effective RSS
  Other Names: Repetitive somatosensory stimulation (RSS); Sham Repetitive somatosensory stimulation (RSS)

SUMMARY:
The study is a comparative study, to show that the administration of RSS stimulation on the face compared to the administration of strategy Sham stimulation, results in an temporary improvement in the tactile acuity of the hand in patients with tactile acuity impairment of the hand due to stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age: 30-80 years old
* Patients with diagnosis of unilateral (both right and left) ischemic or haemorrhagic stroke
* Stroke event dates at least 3 months before the date of inclusion to the study
* Mild-to-moderate sensory loss at the fingers of the hand contralateral to the stroke lesion (affected hand)
* Capacity to provide written consent
* Affiliation to a social security scheme

Non-Inclusion Criteria:

* Sensory impairment attributable to diabetes history, peripheral vascular disease or neuropathy
* Severe speech disorder, global aphasia and/or cognitive impairment
* Multiple stroke events
* Bilateral stroke event
* Hemineglect
* History of neurological or psychiatric illness
* Allergy to glue/tape
* Male participants refusing to shave their moustaches or beards during the study
* Other experimental procedure is forbidden during the weeks where the study is performed
* Pregnant, parturient and lactating women
* Persons deprived of their liberty
* Adult persons subject to a legal protection measure: guardianship, curatorship
* Congenital or acquired malformation/injury of the test finger

Exclusion Criteria:

* Impossibility to maintain hand position necessary for the tests due to severe spasticity
* Severe impairment of the sensibility of the face preventing the administration of the RSS
* Severe impairment of the absolute touch detection at the affected hand preventing measurement (threshold 512 mN)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2023-02-21 (Estimated)

PRIMARY OUTCOMES:
Tactile acuity : 2 point discrimination test | Week 3
  The Primary outcome measure is a composite of 2point discrimination test (2PDT) and Absolute threshold detection test after 3h of RSS.
  Spatial discrimination of the finger, Absolute threshold detection of the finger.
Tactile acuity : Absolute threshold detection test after 3h of RSS | Week 3
  The Primary outcome measure is a composite of 2point discrimination test (2PDT) and Absolute threshold detection test after 3h of RSS.
  Spatial discrimination of the finger, Absolute threshold detection of the finger.

SECONDARY OUTCOMES:
Jebsen-Taylor hand function test (JTHFT) | Week 3
  Overall functionality of the hand, especially with regard to handling objects
Questionnaire comfort/ease to use | Week 3
  A self-reported assessment will be administered after the completion of testing procedure: a custom-made questionnaire including the ease of use, perceived sensations during RSS, easy positioning, pain on removal, positive and negative aspects of RSS, willing to continue using after release from the hospital, and willing to recommend to others.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques LUAUTE, PU-PH, Principal Investigator — Service de Médecine Physique et Réadaptation
Locations (1):
- Groupement Hospitalier du Sud - Hôpital Henry Gabrielle, Saint-Genis-Laval, France